CLINICAL TRIAL: NCT05933980
Title: Combination of Regorafenib，Toripalimab and Celecoxib in Mismatch Repair (MMR) Proficient Refractory Advanced Colorectal Cancer Without Liver Metastasis：a Single Arm Phase II REGOTORICOX Study.
Brief Title: Toripalimab,Celecoxib and Regorafenib in the Treatment of Refractory Advanced Colorectal Cancer
Acronym: REGOTORICOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, professor;chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU26
Record Dates: First submitted 2023-06-24; First posted 2023-07-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Liver Metastases; MSS
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- regorafenib,Toripalima and celecoxib (Experimental): Regorafenib:in dose ramping stage,the initial dose is 80mg per dose, taken orally once a day. After 3 weeks of treatment, the medication is stopped for 1 week (i.e. from day 1 to day 21 and not from day 22 to day 28), with a treatment cycle of 4 weeks.The optimal recommended dose of regofinib (80mg, 120mg, or 160mg) obtained from the phase Ib dose ramping was included in the phase II study dose extension queue.
  Toripalimab:240mg, intravenous drip, administered every three weeks. celecoxib:200mg each time, taken orally twice a day.
  Interventions: Drug: Rego+Tori+Cele

INTERVENTIONS:
Drug: Rego+Tori+Cele — combination of Toripalimab,regorafenib and celecoxib
  Other Names: Bayer AG; Innovent Biologics

SUMMARY:
Research has found that patients with microsatellite instability (dMMR/MSI-H) type colorectal cancer can achieve long-term survival through immune checkpoint inhibitors (ICIs) treatment, but currently accounting for about 95% of MSS type mCRC, the benefits from immune checkpoint inhibitors are very limited. REGONIVO is a Phase Ib study to explore the efficacy and safety of regorafenib in combination with nivolumab in the treatment of gastric cancer and colorectal cancer with MSS. The study enrolled 50 patients with advanced disease, including 25 cases of gastric cancer, 25 cases of colorectal cancer, except for one case of colorectal cancer with MSI-H, and others were MSS type. The results of the study showed that patients with colorectal cancer had an objective response rate (ORR) of 36%.The ORR of liver matestasis vs. lung matestasis is 8.7% vs. 50%.

In this study, pMMR /MSS type patients with refractory advanced colorectal cancer without liver metastasis were selected as the subjects. Regorafenib, Toripalimab and Celecoxib were used to evaluate the maximum tolerable dose, objective response rate (ORR), total survival time (OS), progression free survival time (PFS), disease control rate (DCR), response duration (DoR) and safety of the subjects.

DETAILED DESCRIPTION:
At present, the microsatellite stabilized (MSS) type of advanced refractory metastatic colorectal cancer (mCRC) has a poor median overall survival time of only about 7 months, and there is a significant unmet clinical demand for the efficacy of posterior treatment. Research has found that patients with microsatellite instability (dMMR/MSI-H) type colorectal cancer can achieve long-term survival through immune checkpoint inhibitors (ICIs) treatment, but currently accounting for about 95% of MSS type mCRC, the benefits from immune checkpoint inhibitors are very limited. REGONIVO is a Phase Ib study to explore the efficacy and safety of regorafenib in combination with nivolumab in the treatment of gastric cancer and colorectal cancer with MSS. The study enrolled 50 patients with advanced disease, including 25 cases of gastric cancer, 25 cases of colorectal cancer, except for one case of colorectal cancer with MSI-H, and others were MSS type. The results of the study showed that patients with colorectal cancer had an objective response rate (ORR) of 36%.The ORR of liver matestasis vs. lung matestasis is 8.7% vs. 50%.A phase Ib /Ⅱ clinical study REGOTORI enrolled 39 subjects, with a total ORR of 15.2%, and the ORR of non-liver metastasis subjects compared with liver metastasis subjects was 30% and 8.7% respectively. Based on the prospective small sample clinical trial results of other regifenib combined with PD-1 monoclonal antibody drugs, the overall ORR is between 0% and 33.3%, the ORR for non-liver metastases is between 20% and 50%, and the ORR for liver metastases is between 0% and 15%.

In this study, pMMR /MSS type patients with refractory advanced colorectal cancer without liver metastasis were selected as the subjects. Regorafenib, Toripalimab and Celecoxib were used to evaluate the maximum tolerable dose, objective response rate (ORR), total survival time (OS), progression free survival time (PFS), disease control rate (DCR), response duration (DoR) and safety of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. With subject's consent and signed informed consent form, willing and capable of following planned visits, research treatments, laboratory tests, and other trial procedures
2. Subjects diagnosed with colon or rectal adenocarcinoma by pathology or cytology have evidence of locally advanced lesions or metastases that cannot be surgically removed, without liver metastasis, and all other histological types are excluded.
3. Age 18 and above.
4. The subject has received at least second-line standard chemotherapy in the past and has failed. These standard treatment protocols must include fluorouracil, Oxaliplatin, irinotecan, and Bevacizumab. Subjects with left colon cancer RAS/BRAF V600E genotype of wild type must have received Cetuximab or Panitumumab and other Epidermal growth factor receptor inhibitors. The definition of treatment failure is: disease progression or intolerable toxic side effects occur during the treatment process or within 3 months after the last treatment (One or more chemotherapy drugs with a duration of ≥ 1 cycle for each frontline treatment until the disease progresses; adjuvant/neoadjuvant treatment is allowed in the early stage. If there is recurrence or metastasis during the adjuvant/neoadjuvant treatment or within 6 months after completion, adjuvant/neoadjuvant treatment is considered a failure of frontline systemic chemotherapy for advanced diseases.
5. The Eastern Cancer Cooperative Group's Physical Fitness Score (ECOG) is 0-1 points.
6. Clearly identify measurable lesions that meet the requirements of the evaluation criteria for solid tumor efficacy (RECIST version 1.1)
7. Based on the following laboratory test values obtained during the screening period, appropriate organ function is achieved: white blood cell count ≥ 3.3 × 109/L, neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 75 × 109/L, serum total bilirubin ≤ 1.5 × Upper limit of normal value (UNL), Aspartate transaminase or alanine aminotransferase ≤ 2.5 × UNL (liver metastasis subjects should be ≤ 5 × ULN), serum creatinine ≤ 1.5 × UNL.
8. Female subjects of childbearing age must carry out a serum Pregnancy test within 3 days before starting the study medication, and the result is negative, and are willing to use a medically approved effective contraceptive measure (such as Intrauterine device, contraceptives or condoms) during the study period and within 3 months after the last administration of the study medication.For male subjects whose partners are women of childbearing age, they should undergo surgical sterilization or agree to use effective methods of contraception during the study period and within 3 months after the last study administration.

Exclusion Criteria:

1. Previous or concurrent existence of other active malignant tumors (except malignant tumors that have received cured therapy and have not developed for more than 5 years or Carcinoma in situ that can be cured through adequate treatment);
2. At present, there are duodenal ulcer, Ulcerative colitis, Bowel obstruction and other digestive tract diseases or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers.
3. Thrombosis or embolism events occurred within 6 months before the study, such as cerebrovascular accident (including transient ischemic attack), Pulmonary embolism, Deep vein thrombosis.
4. Within the 6 months prior to enrollment in the study, the following conditions occurred: myocardial infarction, severe/unstable angina, NYHA grade 2 or above cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmias, and symptomatic congestive heart failure.
5. Systemic use of antibiotics for ≥ 7 days within 4 weeks prior to enrollment in the study, or unexplained fever >38.5°C occurring during the screening period/before the first administration (according to the investigator's judgment, fever caused by tumor can be enrolled).
6. Major operations such as laparotomy, thoracotomy, organ removal through Laparoscopy or severe trauma were performed within 4 weeks before the study (Surgical incision should be completely healed before randomization);
7. Within 7 days prior to enrollment in the study, there were uncontrollable pleural effusion, ascites, or pericardial effusion after effective treatment.
8. Immunosuppressive drugs were used within 7 days before the enrollment study, excluding nasal and inhaled Corticosteroid or systemic Sex hormone hormones with physiological dose (i.e. no more than 10mg /d prednisone or other Corticosteroid with physiological dose of equivalent drugs).
9. The general term standard for adverse events (NCICTCAE Version 5.0) caused by any previous treatment that has not yet subsided has toxicity of grade 2 or above (except anemia, hair loss, skin pigmentation and peripheral neurotoxicity related to Oxaliplatin).
10. There are any active, known or suspected autoimmune diseases. Subjects who were in a stable state at the time of enrollment and did not need systemic immunosuppression treatment, such as type I diabetes, hypothyroidism only requiring hormone replacement treatment, and skin diseases that did not need systemic treatment (such as Vitiligo, psoriasis, and alopecia) are allowed.
11. There are Interstitial lung disease, non infectious pneumonia or uncontrollable systemic diseases (such as diabetes, hypertension, Pulmonary fibrosis and acute pneumonia).
12. HIV (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; hepatitis C, defined as HCV-RNA higher than the detection limit of the analytical method) or co infection of hepatitis B and C.
13. Previously received antibodies against Programmed cell death protein-1 (PD-1) or its ligand (PD-L1), antibodies against cytotoxic T-lymphocyte associated protein 4 (CTLA-4), or other drugs/antibodies that act on the costimulation or checkpoint pathway of T cells.
14. Previous treatment with regofinib.
15. Medical history of known or suspected allergy to any relevant Drug allergy used in the study.
16. Pregnant or lactating women.
17. Women of childbearing age who have not used or refused to use effective non hormonal contraceptive methods (<2 years after their last menstrual period) or men who are at risk of giving birth.
18. The presence of other serious physical or mental illnesses or laboratory examination abnormalities may increase the risk of participating in the study, or interfere with the results of the study, as well as subjects deemed unsuitable by the researcher for participation in this study。

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 years
  objective response rate

SECONDARY OUTCOMES:
OS | 2 years
  total survival time
PFS | 2 years
  progression free survival time
DCR | 2 years
  disease control rate
DoR | 2 years
  response duration

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, docter, Principal Investigator — The Six Affiliated Hospital,Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Akin Telli T, Bregni G, Vanhooren M, Saude Conde R, Hendlisz A, Sclafani F. Regorafenib in combination with immune checkpoint inhibitors for mismatch repair proficient (pMMR)/microsatellite stable (MSS) colorectal cancer. Cancer Treat Rev. 2022 Nov;110:102460. doi: 10.1016/j.ctrv.2022.102460. Epub 2022 Aug 27. PMID 36058142
- [Background] Andre T, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Bendell J, Le DT, Yoshino T, Van Cutsem E, Yang P, Farooqui MZH, Marinello P, Diaz LA Jr; KEYNOTE-177 Investigators. Pembrolizumab in Microsatellite-Instability-High Advanced Colorectal Cancer. N Engl J Med. 2020 Dec 3;383(23):2207-2218. doi: 10.1056/NEJMoa2017699. PMID 33264544
- [Background] Fukuoka S, Hara H, Takahashi N, Kojima T, Kawazoe A, Asayama M, Yoshii T, Kotani D, Tamura H, Mikamoto Y, Hirano N, Wakabayashi M, Nomura S, Sato A, Kuwata T, Togashi Y, Nishikawa H, Shitara K. Regorafenib Plus Nivolumab in Patients With Advanced Gastric or Colorectal Cancer: An Open-Label, Dose-Escalation, and Dose-Expansion Phase Ib Trial (REGONIVO, EPOC1603). J Clin Oncol. 2020 Jun 20;38(18):2053-2061. doi: 10.1200/JCO.19.03296. Epub 2020 Apr 28. PMID 32343640
- [Background] Wang F, He MM, Yao YC, Zhao X, Wang ZQ, Jin Y, Luo HY, Li JB, Wang FH, Qiu MZ, Lv ZD, Wang DS, Li YH, Zhang DS, Xu RH. Regorafenib plus toripalimab in patients with metastatic colorectal cancer: a phase Ib/II clinical trial and gut microbiome analysis. Cell Rep Med. 2021 Aug 27;2(9):100383. doi: 10.1016/j.xcrm.2021.100383. eCollection 2021 Sep 21. PMID 34622226